CLINICAL TRIAL: NCT02440932
Title: Impact of Phenylketonuria-type Diet on Appetite, Appetite Hormones and Diet Induced Thermogenesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Dr Dalia Malkova, Senior Lecturer, University of Glasgow
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 200130139
Record Dates: First submitted 2015-04-30; First posted 2015-05-12 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Phenylketonuria (PKU)
Keywords: low Phenylalanine diet; PKU supplements; diet induced thermogenesis; appetite; body weight
MeSH Terms: conditions — Phenylketonurias; Body Weight | interventions — Diet

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phenylketonuria-type diet (Experimental): Breakfast: one pouch of amino acid supplement (174 mls supplemented drink PKU cooler 20, Vitaflo®; 20 g protein, 9.4 g carbohydrates, 0.7 g Fat) Lunch: cheese sandwich [low protein bread (Juvela, UK), no protein vegan cheese (Viotros, UK)], low protein crackers (Vitaflo, UK), and low protein cookies (Juvela, UK).
  Dinner: ad libitum buffet meal
  Interventions: Dietary Supplement: Phenylketonuria-type diet; Other: Normal (control) diet
- Normal diet (Other): Breakfast: 174 ml of milk (20 g protein, 9.4 g carbohydrates, 0.7 g Fat) Lunch: cheese sandwich, crackers, and cookies (regular foods) Dinner: ad libitum buffet meal
  Interventions: Dietary Supplement: Phenylketonuria-type diet; Other: Normal (control) diet

INTERVENTIONS:
Dietary Supplement: Phenylketonuria-type diet — Breakfast, lunch and open buffet dinner
Other: Normal (control) diet — Breakfast, lunch and open buffet dinner

SUMMARY:
Low-phenylalanine diets are commonly prescribed to people with phenylketonuria (PKU), an inborn disease which causes accumulation of amino acid phenylalanine (Phe) in the blood. High blood Phe levels can cause mental, behavioural, neurological, and physical problems. Thus, low-phenylalanine diets help patients to manage their condition but it is not clear whether they have an impact on appetite, energy intake and changes in body weight. This is important to explore as prevalence of obesity in this population is rising high. This study aims to find out the effect of PKU-type meals on appetite, appetite biomarkers, and post-meal energy expenditure. The investigators will recruit 26 healthy adults and ask them to participate in two experimental trials. On one occasion the participants will be asked to consume a PKU-supplemented drink followed by a PKU type-lunch and on another occasion the supplement and lunch will be based on normally consumed foods. Series of blood samples will be taken and appetite will be assessed during both experiments. Both experimental trials will finish with consuming an "all-you-can-eat" buffet.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult
2. Body weight stable for previous 4 months
3. Regular menstrual cycle (females)

Exclusion Criteria:

1. Pregnancy or lactation (females)
2. History of eating disorder
3. History of gastrointestinal problems or surgery
4. History of allergy
5. History of chronic illness
6. On any medication
7. Smoking
8. On nutritional supplements
9. Following specific diet
10. Currently taking part in other research

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2014-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Appetite hormone: peptide YY (PYY) | 300 minutes
  Plasma concentration at baseline (0 minute) and after ingestion of supplement (at 30, 60 and 90 minutes) and lunch (at 120, 150,180, 210, 240, 270 and 300 minutes)
Appetite hormone: glucagon-like peptide-1 (GLP-1) | 300 minutes
  Plasma concentration at baseline (0 minute) and after ingestion of supplement (at 30, 60 and 90 minutes) and lunch (at 120, 150,180, 210, 240, 270 and 300 minutes)
Appetite hormone: cholecystokinin (CCK) | 300 minutes
  Plasma concentration at baseline (0 minute) and after ingestion of supplement (at 30, 60 and 90 minutes) and lunch (at 120, 150,180, 210, 240, 270 and 300 minutes)
Appetite hormone: insulin | 300 minutes
  Plasma concentration at baseline (0 minute) and after ingestion of supplement (at 30, 60 and 90 minutes) and lunch (at 120, 150,180, 210, 240, 270 and 300 minutes)
Appetite hormone: ghrelin | 300 minutes
  Plasma concentration at baseline (0 minute) and after ingestion of supplement (at 30, 60 and 90 minutes) and lunch (at 120, 150,180, 210, 240, 270 and 300 minutes)
Subjective appetite score | 300 minutes
  Visual analogue scale (VAS) collected at baseline and after each blood sample collection
Diet induced thermogenesis | 300 minutes
  Metabolic rate by means of computerised open-circuit ventilated hood system collected at baseline and after each blood sample collection for the duration of 20 minutes

SECONDARY OUTCOMES:
Taste perception of PKU supplements/foods | 10 minutes
  Immediately after supplement ingestion and lunch consumption
Consumption time for PKU supplements/foods | 20 minutes
  Maximum 5 minutes for supplement ingestion and maximum 20 minutes for lunch consumption

CONTACTS AND LOCATIONS:
Overall Officials: Dalia Malkova, PhD, Study Chair — University of Glasgow
Locations (1):
- Human Nutrition, School of Medicine, University of Glasgow, Glasgow, United Kingdom

REFERENCES:
- [Derived] Alfheeaid H, Gerasimidis K, Nastase AM, Elhauge M, Cochrane B, Malkova D. Impact of phenylketonuria type meal on appetite, thermic effect of feeding and postprandial fat oxidation. Clin Nutr. 2018 Jun;37(3):851-857. doi: 10.1016/j.clnu.2017.03.005. Epub 2017 Mar 8. PMID 28318688